CLINICAL TRIAL: NCT03139227
Title: Celery-Based Dietary Intervention: A Feasibility Study
Brief Title: Apigenin in Increasing Health Benefits in High Risk Breast Clinic Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI decision
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Sagar Sardesai, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-17006; NCI-2017-00517 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2017-04-17; First posted 2017-05-03 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Health Status Unknown
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (celery-banana bread) (Experimental): Patients consume one serving of lower dose apigenin celery-banana bread daily on days 1-7, and then consume one serving of higher dose apigenin celery-banana bread on days 8-14. Patients undergo blood sample collection on day 1 prior to and 6 hours after bread ingestion, on day 8 prior to and 6 hours after ingestion of bread, and on day 15 (or endpoint). Patients also provide a baseline urine sample and then 24-hour urine samples on days 1, 7, 8, and 14.
  Interventions: Procedure: Bio specimen Collection; Dietary Supplement: Dietary Intervention; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Procedure: Bio specimen Collection — Patients undergo collection of blood and urine
Dietary Supplement: Dietary Intervention — Consume celery-banana bread
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies the side effects and best dose of apigenin in increasing health benefits in high risk breast clinic patients. Celery is high in apigenin, a compound that may have anti-cancer activities. Eating a celery-based diet may help in prevention and treatment of inflammatory diseases including cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES; I. To determine the feasibility of apigenin oral supplementation using a specially formulated celery-banana bread.

II. To determine the safety and tolerability of apigenin supplementation.

OUTLINE: This is a dose-escalation study.

Patients consume one serving of lower dose apigenin celery-banana bread daily on days 1-7, and then consume one serving of higher dose apigenin celery-banana bread on days 8-14. Patients undergo blood sample collection on day 1 prior to and 6 hours after bread ingestion, on day 8 prior to and 6 hours after ingestion of bread, and on day 15 (or endpoint). Patients also provide a baseline urine sample and then 24-hour urine samples on days 1, 7, 8, and 14.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be followed in Stefanie Spielman Comprehensive Breast Center (SSCBC) High Risk Breast Clinic
* No known allergy to ingredients of banana bread preparation (eggs, almonds and other nuts since the celery also has almond powder)
* Must be > 1 year from pregnancy, lactation or chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Ability to give informed consent
* Participate in the specified study visits and laboratory testing including three (20 mL) blood draws and three 24 hour urine collections

Exclusion Criteria:

* Concurrent malignancy or metastatic malignancy of any kind
* Ongoing chemotherapy, radiation therapy, or other cancer-related treatment
* Current and past history of hypertension
* Chronic use of any herbal or dietary supplement containing apigenin within the 3 months prior to entry on the study
* Pregnant or nursing women
* Concurrent use of tamoxifen, raloxifene, or any of the aromatase inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-03-14 (Actual)

PRIMARY OUTCOMES:
Apigenin levels in blood and urine | Up to 14 days
  Paired t-tests will be used to compare mean apigenin levels.

CONTACTS AND LOCATIONS:
Overall Officials: Sagar Sardesai, MBBS, Principal Investigator — Ohio State University Comprehensive Cancer Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu